CLINICAL TRIAL: NCT03626857
Title: MiACLR: Michigan Initiative for Anterior Cruciate Ligament Rehabilitation
Acronym: MiACLR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Connecticut (Other); University of Delaware (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Riann Palmieri-Smith, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00144992; 1R01HD093626-01A1 (NIH)
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Results first posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: Knee; ACL; Reconstruction; Rehabilitation; Eccentric Exercise; Electrical Stimulation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMES+ECC (Experimental): Neuromuscular electrical stimulation (NMES) and Eccentric Exercise (ECC). Patients randomized to the NMES+ECC group will first receive NMES for 2x/week for 8 weeks, beginning at the first post-operative visit. Beginning at 9 weeks after anterior cruciate ligament reconstruction (ACLR) patients will begin to receive eccentric exercise 2x/week for an additional 8 weeks. For NMES, patients will have electrical stimulation delivered to their quadriceps. Fifteen isometric actions lasting 10 seconds each will be elicited during each session. For eccentric exercise, patients will train for 4 sets of 10 repetitions. This group will also receive standard of care ACL rehabilitation alongside the study interventions.
  Interventions: Device: Neuromuscular Electrical Stimulation (NMES); Other: Eccentric Exercise (ECC)
- NMES placebo + ECC placebo (Placebo Comparator): Neuromuscular electrical stimulation (NMES) low intensity/placebo + Eccentric Exercise (ECC) low intensity/placebo arm. Patients randomized to the NMES low intesntiy/placebo + ECC low intensity/placebo group will first receive NMES placebo/low-intensity treatment for 2x/week for 8 weeks, beginning at the first post-operative physical therapy visit. Beginning at 9 weeks after anterior cruciate ligament reconstruction (ACLR) patients will begin to receive an eccentric exercise low-intensity/placebo 2x/week for 8 weeks.
  For the NMES low intensity/placebo, patients will have it delivered to their quadriceps 2x/week for 8 weeks beginning at the first post-operative visit. Fifteen isometric actions lasting 10 seconds each will be elicited during each session.
  For the eccentric exercise low-intensity/placebo, patients will begin to receive eccentric exercise two times per week for 8 weeks. Patients will train for 4 sets of 10 repetitions.
  Interventions: Device: Neuromuscular Electrical Stimulation (NMES) placebo; Other: Eccentric Exercise (ECC) placebo

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation (NMES) — The electrical stimulator will deliver a 2500 Hz alternating current, modulated at 75 bursts/s, with a ramp-up time of 2-seconds, followed by a 50-second rest period. Stimulus intensity set to generate a maximum voluntary isometric contraction (MVIC) of at least 40& of the contralateral MVIC.
  Other Names: Electrical Stimulation; Estim
  Arms: NMES+ECC
Other: Eccentric Exercise (ECC) — 4 sets of 10 repetitions of an eccentric leg press exercise performed at 70-90% of the 1 repetition maximum
  Arms: NMES+ECC
Device: Neuromuscular Electrical Stimulation (NMES) placebo — The electrical stimulator will deliver a 2500 Hz alternating current, modulated at 75 bursts/s, with a ramp-up time of 2-seconds, followed by a 50-second rest period. Stimulus intensity set to generate a maximum voluntary isometric contraction (MVIC) of 10-20% of the contralateral MVIC.
  Arms: NMES placebo + ECC placebo
Other: Eccentric Exercise (ECC) placebo — 4 sets of 10 repetitions of an eccentric leg press exercise performed at 10-20% of the 1 repetition maximum
  Arms: NMES placebo + ECC placebo

SUMMARY:
This clinical trial evaluates interventions to maximize muscle function and improve cartilage health following anterior cruciate ligament reconstruction. Improving muscle function may improve patient outcomes, improve joint mechanics, and potentially serve as a prevention approach for post-traumatic knee osteoarthritis. Knee osteoarthritis (OA) is a disabling disease that carries a substantial burden to society and to the individual affected.

DETAILED DESCRIPTION:
Restoring quadriceps muscle strength following anterior cruciate ligament reconstruction (ACLR) may help prevent the post-traumatic knee osteoarthritis that affects over 50% of knees 10-20 years after surgical reconstruction. However, a fundamental gap exists in current understanding of how to maximize muscle strength following ACLR, as current rehabilitation fails to restore symmetrical quadriceps strength. The investigators pilot work shows that when patients return to activity, quadriceps strength is ~70% of the uninjured side, which is far below the recommended 90%. Further, these data suggest that embedding high-intensity neuromuscular electrical stimulation (NMES) and eccentric exercise into standard of care ACL rehabilitation leads to higher quadriceps strength when compared with standard of care alone. However, the true efficacy of these interventions is unknown, as controlled trials with adequate sample sizes are currently lacking. The absence of this information serves as the driving force and focus of the proposed trial. Therefore, the investigators propose a double-blind randomized controlled trial where ACLR patients will be randomized to 1 of 2 arms. Study arms will include: 1) 8 weeks of NMES+8 weeks of eccentric exercise; 2) 8 weeks of NMES placebo+8 weeks of eccentric placebo. All study arms will receive standard of care ACL rehabilitation in addition to the study interventions. The investigators hypothesize that subjects receiving NMES+eccentric exercise (Arm 1) will realize greater improvements in strength and biomechanical function at 6 months following ACLR than patients in the placebo study arm. Further, the investigators anticipate that patients in the NMES+eccentric exercise arm (Arm 1) will best eliminate negative changes in cartilage health at 18 months following ACLR. This study is innovative, because it employs interventions that directly target the primary mechanisms that result in strength loss following ACLR and will also evaluate whether improving muscle strength can minimize early changes in cartilage health, which may be indicative of future osteoarthritis. The proposed research is significant because it will identify evidence-based treatment approaches that can successfully counteract the muscle weakness which plagues ACLR patients for years after injury and contributes to the onset of post-traumatic osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Acute, complete ACL rupture
* ACL reconstruction with autograft
* Scheduled to undergo ACLR at U of Michigan
* Willingness to participate in testing and follow-up as outlined

Exclusion Criteria:

* Previous surgery to either knee
* Bony fracture accompanying ACL injury
* Patients who experienced a knee dislocation
* Female participants who are pregnant or planning pregnancy

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 135 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - MedSport, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez K, Garcia SA, Spino C, Lepley LK, Pang Y, Wojtys E, Bedi A, Angelini M, Ruffino B, Bolley T, Block C, Kellum J, Swartout A, Palmieri-Smith RM. Michigan Initiative for Anterior Cruciate Ligament Rehabilitation (MiACLR): A Protocol for a Randomized Clinical Trial. Phys Ther. 2020 Dec 7;100(12):2154-2164. doi: 10.1093/ptj/pzaa169. PMID 32939539

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited beginning in January of 2019 through July of 2023 from Michigan Medicine.
Pre-assignment Details: Participants were not randomized after enrollment for the following reasons:
  1. Withdrew Consent
  2. Screen fail
  3. COVID drops (COVID pandemic prevented testing)
  4. Lost to follow-up
  A baseline testing session occurred prior to randomization.
Groups:
- Active High-Intensity NMES+ECC: Neuromuscular electrical stimulation (NMES) and Eccentric Exercise (ECC). Patients randomized to the NMES+ECC group will first receive high-intensity NMES for 2x/week for 8 weeks, beginning at the first post-operative visit. Beginning approximately 9 weeks after anterior cruciate ligament reconstruction (ACLR) patients will begin to receive eccentric exercise 2x/week for an additional 8 weeks. For NMES, patients will have electrical stimulation delivered to their quadriceps. Fifteen isometric actions lasting 10 seconds each will be elicited during each session. For eccentric exercise, patients will train for 4 sets of 10 repetitions. This group will also receive standard of care ACL rehabilitation alongside the study interventions.
- Placebo Low-Intensity NMES + ECC: Neuromuscular electrical stimulation (NMES) low intensity/placebo + Eccentric Exercise (ECC) low intensity/placebo arm. Patients randomized to the NMES low intesntiy/placebo + ECC low intensity/placebo group will first receive NMES placebo/low-intensity treatment for 2x/week for 8 weeks, beginning at the first post-operative physical therapy visit. Beginning at 9 weeks after anterior cruciate ligament reconstruction (ACLR) patients will begin to receive an eccentric exercise low-intensity/placebo 2x/week for 8 weeks.
  For the NMES low intensity/placebo, patients will have it delivered to their quadriceps 2x/week for 8 weeks beginning at the first post-operative visit. Fifteen isometric actions lasting 10 seconds each will be elicited during each session.
  For the eccentric exercise low-intensity/placebo, patients will begin to receive low dose eccentric exercise two times per week for 8 weeks. Patients will train for 4 sets of 10 repetitions.
Period: Overall Study
Arm/Group | Active High-Intensity NMES+ECC | Placebo Low-Intensity NMES + ECC
Started | 57 | 56
Post-NMES Intervention Testing | 53 | 53
Post-ECC Intervention Testing | 52 | 50
9 month post-ACLR testing | 49 | 44
18 month post-ACLR testing | 37 | 36
Completed | 37 | 36
Not Completed | 20 | 20
Not completed — Adverse Event | 9 | 7
Not completed — Lost to Follow-up | 8 | 8
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NMES+ECC | NMES Placebo + ECC Placebo | Total
Number analyzed (Participants) | 57 | 56 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.9 (7.1) | 23.0 (8.1) | 22.9 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 31 | 30 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 8 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 10 | 17
  White | 40 | 36 | 76
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 54 | 51 | 105
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Immediately Post NMES+ECC Intervention Isokinetic Quadriceps Strength Index
Description: Bilateral concentric isokinetic muscle strength at 60 degrees per second. Limb symmetry index is calculated as (ACL strength/Non-ACL strength)*100
Time Frame: Post-NMES+ECC intervention (approximately 16 weeks post-ACL reconstruction)
Population: Active High-Intensity NMES + ECC: 2 subjects withdrawn by investigator, 0 subjects lost to follow up, 1 subject withdrew consent, 2 people missing strength data Placebo Low-Intensity NMES + ECC: 1 subjects withdrawn by investigator, 2 subjects lost to follow up, 2 subject withdrew consent, 1 person missing strength data
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | NMES+ECC | NMES placebo + ECC placebo
Number analyzed (Participants) | 52 | 50
Percentage | 60.9 (20.5) | 58.4 (19.2)
Statistical Analysis 1: Comparison: NMES+ECC vs NMES placebo + ECC placebo; Test type: Superiority; p = .025, Mixed Models Analysis

2. Primary Outcome: 9 Months Isokinetic Quadriceps Strength Limb Symmetry Index
Description: as for outcome 1
Time Frame: 9 months (9 months post-ACL reconstruction)
Population: Active High-Intensity NMES + ECC: 3 subjects withdrawn by investigator, 4 subjects lost to follow up, 1 subject withdrew consent Placebo Low-Intensity NMES + ECC: 4 subjects withdrawn by investigator, 6 subjects lost to follow up, 2 subject withdrew consent
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | NMES+ECC | NMES placebo + ECC placebo
Number analyzed (Participants) | 49 | 44
Percentage | 76.8 (18.0) | 74.5 (19.6)
Statistical Analysis 1: Comparison: NMES+ECC vs NMES placebo + ECC placebo; Test type: Superiority; p = 0.025, Mixed Models Analysis

3. Secondary Outcome: Knee Flexion Angle at 9 Months
Description: Peak knee flexion angle of the ACL leg recorded during a single-legged hop (units: degrees)
Time Frame: 9 months post-ACL reconstruction
Population: Active High-Intensity NMES + ECC : 3 subjects withdrawn by investigator, 4 subjects lost to follow up, 1 subject withdrew consent, 16 subjects could not complete a single leg hop so data is missing Placebo Low-Intensity NMES + ECC: 4 subjects withdrawn by investigator, 6 subjects lost to follow up, 2 subject withdrew consent, 10 subjects could not complete a single leg hop so data is missing
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | NMES+ECC | NMES placebo + ECC placebo
Number analyzed (Participants) | 33 | 34
Degrees | 50.9 (14.4) | 44.4 (12.9)

4. Secondary Outcome: Knee Flexion Moment at 9 Months
Description: Peak knee flexion moment recorded during a single-legged hop (units: Nm/kg*m)
Time Frame: 9 months post-ACL reconstruction
Population: Active High-Intensity NMES + ECC: 3 subjects withdrawn by investigator, 4 subjects lost to follow up, 1 subject withdrew consent, 16 subjects could not complete a single leg hop so data is missing Placebo Low-Intensity NMES + ECC: 4 subjects withdrawn by investigator, 6 subjects lost to follow up, 2 subject withdrew consent, 10 subjects could not complete a single leg hop so data is missing
Measure: Mean (Standard Deviation); unit: Nm/kg*m
Arm/Group | NMES+ECC | NMES placebo + ECC placebo
Number analyzed (Participants) | 33 | 34
Nm/kg*m | 1.4 (0.3) | 1.3 (0.3)

5. Secondary Outcome: Knee Flexion Angle at 18 Months
Description: Peak knee flexion angle recorded during a single-legged hop (units: degrees)
Time Frame: 18 months post-ACL reconstruction
Population: Active High-Intensity NMES + ECC: 10 subjects withdrawn by investigator, 8 subjects lost to follow up, 2 subjects withdrew consent, 7 subjects could not complete a single leg hop so data is missing Placebo Low-Intensity NMES + ECC: 7 subjects withdrawn by investigator, 10 subjects lost to follow up, 2 subjects withdrew consent, 6 subjects could not complete a single leg hop so data is missing
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | NMES+ECC | NMES placebo + ECC placebo
Number analyzed (Participants) | 30 | 31
Degrees | 53.4 (14.7) | 48.8 (11.4)

6. Secondary Outcome: Knee Flexion Moment at 18 Months
Description: Peak knee flexion moment recorded during a single-legged hop (units: Nm/kg*m)
Time Frame: 18 months post-ACL reconstruction
Population: Active High-Intensity NMES + ECC: 10 subjects withdrawn by investigator, 8 subjects lost to follow up, 2 subject withdrew consent, 7 subjects could not complete a single leg hop so data is missing Placebo Low-Intensity NMES + ECC: 7 subjects withdrawn by investigator, 10 subjects lost to follow up, 2 subject withdrew consent, 6 subjects could not complete a single leg hop so data is missing
Measure: Mean (Standard Deviation); unit: Nm/kg*m
Arm/Group | NMES+ECC | NMES placebo + ECC placebo
Number analyzed (Participants) | 30 | 31
Nm/kg*m | 1.5 (0.4) | 1.5 (0.3)

7. Secondary Outcome: T1 Rho Relaxation Time Symmetry Score for Femoral Knee Joint Cartilage
Description: [T1rho value at the weight bearing region of medial femur from MRI for ACL knee (msec)/T1rho value at the weight bearing region of medial femur for NonACL knee (msec)] x 100
Time Frame: 18 months post-ACL reconstruction
Population: Active High-Intensity NMES + ECC: 10 subjects withdrawn by investigator, 8 subjects lost to follow up, 2 subject withdrew consent, 1 person with MRI scan error so data is missing Placebo Low-Intensity NMES + ECC: 7 subjects withdrawn by investigator, 11 subjects lost to follow up, 2 subject withdrew consent
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | NMES+ECC | NMES placebo + ECC placebo
Number analyzed (Participants) | 36 | 36
Percentage | 103.0 (15.9) | 106.1 (21.9)

8. Secondary Outcome: T2 Relaxation Time Symmetry Score for Femoral Knee Joint Cartilage
Description: [T2 value from MRI at the central weight bearing region of femur for the ACL knee (msec)/T2 value from MRI at the central weight bearing region of femur for the NonACL knee (msec)] x 100
Time Frame: 18 months post-ACL reconstruction
Population: NMES+ECC arm: 10 subjects withdrawn by investigator, 8 subjects lost to follow up, 2 subject withdrew consent, 1 person with MRI scan error so data is missing NMES placebo + ECC placebo arm: 7 subjects withdrawn by investigator, 11 subjects lost to follow up, 2 subject withdrew consent
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | NMES+ECC | NMES placebo + ECC placebo
Number analyzed (Participants) | 36 | 36
Percentage | 101.3 (8.7) | 104.4 (9.8)

ADVERSE EVENTS:
Time Frame: From the time of study enrollment until the last study visit occurring at 18 months after ACL reconstruction
Arm/Group | NMES+ECC | NMES Placebo + ECC Placebo
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/56
Serious Adverse Events (participants affected / at risk) | 8/57 | 6/56
Other Adverse Events (participants affected / at risk) | 2/57 | 3/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NMES+ECC (N=57) | NMES Placebo + ECC Placebo (N=56)
Appendectomy (Surgical and medical procedures) | 1 | 0 — Unrelated to intervention
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0 — Unrelated to Intervention
Septoplasty (Surgical and medical procedures) | 0 | 1 — Unrelated to Intervention
Loss of Consciousness (Nervous system disorders) | 0 | 1 — Unrelated to Intervention
Hospitalization for severe persistent asthma w/ exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Unrelated to Intervention
Meniscal Surgery (Surgical and medical procedures) | 3 | 0 — Unrelated to Intervention
Cyclops lesion excision (Surgical and medical procedures) | 1 | 1 — Unrelated to intervention
Anterolateral Ligament Reconstruction with partial ACL graft tear (Musculoskeletal and connective tissue disorders) | 1 | 0
Contralateral ACL tear (Musculoskeletal and connective tissue disorders) | 1 | 1 — Not related to the intervention
Knee arthroscopy (Musculoskeletal and connective tissue disorders) | 0 | 1 — Not related to the intervention
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NMES+ECC (N=57) | NMES Placebo + ECC Placebo (N=56)
ACL graft tear that was not reconstructed (Musculoskeletal and connective tissue disorders) | 2 | 3 — Not related to intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT03626857/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT03626857/ICF_001.pdf